CLINICAL TRIAL: NCT05288842
Title: TANYCYTES' ROLE IN ALZHEIMER'S DISEASE AND FRONTOTEMPORAL DEMENTIA: ARE THEY THE KEY TO WELL AGING?
Brief Title: Tanycytes in Alzheimer's Disease and Frontotemporal Dementia
Acronym: BIOWATCH
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: European Research Council (Other); CH Calais (Unknown); Centre Hospitalier VALENCIENNES (Other); Région Nord-Pas de Calais, France (Other); Centre Hospitalier de Bethune (Network)
Responsible Party: Sponsor
Other Study IDs: 2020_26; 2021-A00879-32 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2021-07-27; First posted 2022-03-21 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Alzheimer Disease; Frontotemporal Dementia
Keywords: Alzheimer disease; Frontotemporal Dementia; tanycytes; metabolism; hormone; cerebrospinal fluid; blood; hypothalamus
MeSH Terms: conditions — Alzheimer Disease; Frontotemporal Dementia | interventions — Spinal Puncture; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma and CSF supernatant will be aliquoted and labelled for storage
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Controls
  Interventions: Biological: Lumbar puncture; Biological: blood sample
- Group 2: Alzheimer's Disease
  Interventions: Biological: Lumbar puncture; Biological: blood sample
- Group 3: Frontotemporal Dementia
  Interventions: Biological: Lumbar puncture; Biological: blood sample

INTERVENTIONS:
Biological: Lumbar puncture — 5 mL of CSF
Biological: blood sample — 6x5 mL of blood sample collected :1 dry tube, 2 EDTA tubes, 1 fluoride tube, and 2 polypropylene tubes

SUMMARY:
Metabolic and hormonal deregulations are both a risk factor and a hallmark of Alzheimer's disease (AD) and frontotemporal dementia (FTD), occurring early in the course of the disease. In FTD in particular, hyperorality and dietary changes are associated with metabolic and hormonal changes such as altered levels of the anorexigenic hormone leptin.

The hypothalamus is a brain region that controls metabolism and hormonal systems. Hypothalamic function depends on its ability to sense peripheral signals. The hypothalamus sits on a circumventricular organ called the median eminence (ME) that puts it in contact with systemic blood circulation. In the ME, fenestrated capillaries allow the diffusion of bloodborne factors. However, despite the lack of blood-brain barrier at brain microvessels, diffusion is controlled by specialized ependymoglial cells, the tanycytes, which exert a barrier function between the ME and the third ventricle and controls the access of blood-borne molecules into the hypothalamus. Previous work from our laboratory and the ERC consortium has highlighted the role of tanycytes not only in the regulation of the release of neurohormones from neuroendocrine nerve terminals into the pituitary portal blood circulation, but also in the transport of circulating leptin into the hypothalamus. Hence hypothalamic dysfunction in AD and FTD can result either from dysregulation of neuroendocrine secretions, direct neuronal loss or from defective transport (and hence resistance) to hormones like leptin.

This study is to demonstrate that leptin transport though tanycytes is early altered in FTD and AD and correlates

DETAILED DESCRIPTION:
Metabolic and hormonal deregulations are both a risk factor and a hallmark of Alzheimer's disease (AD) and frontotemporal dementia (FTD), occurring early in the course of the disease. In FTD in particular, hyperorality and dietary changes are associated with metabolic and hormonal changes such as altered levels of the anorexigenic hormone leptin.

The hypothalamus is a brain region that controls metabolism and hormonal systems. Hypothalamic function depends on its ability to sense peripheral signals. The hypothalamus sits on a circumventricular organ called the median eminence (ME) that puts it in contact with systemic blood circulation. In the ME, fenestrated capillaries allow the diffusion of bloodborne factors. However, despite the lack of blood-brain barrier at brain microvessels, diffusion is controlled by specialized ependymoglial cells, the tanycytes, which exert a barrier function between the ME and the third ventricle and controls the access of blood-borne molecules into the hypothalamus. Previous work from our laboratory and the ERC consortium has highlighted the role of tanycytes not only in the regulation of the release of neurohormones from neuroendocrine nerve terminals into the pituitary portal blood circulation, but also in the transport of circulating leptin into the hypothalamus. Hence hypothalamic dysfunction in AD and FTD can result either from dysregulation of neuroendocrine secretions, direct neuronal loss or from defective transport (and hence resistance) to hormones like leptin.

Our aim is to demonstrate that leptin transport though tanycytes is early altered in FTD and AD and correlates with metabolic and hormonal alterations, as well as with disease biomarkers.

Moreover, a recent study from our laboratory shows that gonadotropin or GnRH, the hormone that plays an essential role in the survival of our species by controlling the reproductive axis (the hypothalamic-pituitary-gonadal axis, or HPG) from minipuberty (first activation of the HPG after birth occurring as early as the second week of life), to male and female fertility through puberty, also plays a role in cognition and that the alteration of its secretion rate can lead to cognitive decline in certain conditions such as Down's syndrome (T21) and AD. Indeed, our preclinical studies in mouse models of T21 and AD show that an alteration of the pulsatility parameters of GnRH secretion, as evidenced by the alteration of the secretion profile of luteinizing hormone (LH) which is its proxy in the systemic circulation, accompanies cognitive decline and that pharmacological treatment with a subcutaneous pump delivering the natural hormone, GnRH, at the endogenous rate of littermates not carrying TS21 or AD, restores cognitive faculties to levels of mice not carrying the syndrome or the disease. A pilot study on 7 adult patients with T21, shows that the same pulsatile GnRH treatment increases cognition and markedly improves functional connectivity at rest of neuronal circuits known to be impaired in T21 after 6 months of treatment.

We will therefore take benefit of the ongoing BioWATCH study, which assesses hypothalamic function in patients with AD and FTD, to analyze GnRH pulsatility in a subset of participants. The main objective of the UPGRADE ancillary study is to demonstrate that pulsatile GnRH secretion is altered in AD, but also in other dementias such as frontotemporal dementia (FTD), and that this alteration correlates with clinical, imaging or biological markers. We ultimately aim at laying the groundwork for a pulsatile GnRH therapy in AD and FTD.

ELIGIBILITY:
Inclusion Criteria:

* Subjects able to undergo a lumbar puncture
* Subjects registered with the French Social Security, in agreement with the French law on biomedical experimentation

To be assigned in the study subgroups, subjects will have to fulfill the specific following criteria:

Group 1: Controls

* absence of cognitive complaint (completion of the memory complaint questionnaire)
* absence of significant cognitive impairment: normal MMSE according to age and education levels
* Subjects capable of and willing to comply with the protocol and to give their written informed consents after having received and understood the subject information Group 2: Alzheimer's Disease
* Diagnosis of probable Alzheimer's disease dementia according to the NIA 2011 criteria1
* MMSE ≥ 16
* Subjects who have a study partner. The study partner is required to complete several scales and to drive back the subject after the lumbar puncture for safety reasons. If the subjects or their study partners are not able to drive, their transport fees will be reimbursed by the promotor
* Subjects and study partners capable of and willing to comply with the protocol and to give their written informed consents after having received and understood the subject information. According to the legal protection or the mental capacities of the subject, the subject will be accompanied by a legally acceptable representative during this procedure Group 3: Frontotemporal Dementia
* Diagnosis of probable frontotemporal dementia according to the FTDC 2011 criteria2
* MMSE ≥ 16
* Subjects who have a study partner. The study partner is required to complete several scales and to drive back the subject after the lumbar puncture for safety reasons. If the subjects or their study partners are not able to drive, their transport fees will be reimbursed by the promotor
* Subjects and study partners capable of and willing to comply with the protocol and to give their written informed consents after having received and understood the subject information. According to the legal protection or the mental capacities of the subject, the subject be accompanied by a legally acceptable representative during this procedure

Exclusion Criteria:

* General exclusion criteria:
* Subjects with dementia caused by a non-neurodegenerative disease, including patients with severe cerebrovascular risk factor load
* Subjects who have contraindications to perform a lumbar puncture
* Subjects who have contraindications to perform a MRI scan
* Weighted less than 45 kg

Associated illnesses or conditions:

* Subjects with other neurodegenerative disease such as Lewy body dementia and Parkinson's disease
* Subjects with other serious neurological disorder such as brain tumor, stroke, epilepsy, hydrocephalus and any condition which contraindicates, in the investigator's judgment, entry to the study;
* Subjects with severe metabolic or endocrine disorder (excluding hypothyroidism under stable hormone replacement therapy, controlled type 2 diabetes or common dyslipidaemia), previously known or identified at screening
* Subjects under metformin treatment.

Biological exclusion criteria:

* Subjects with known active HCV, HBV or HIV
* Subjects with clinical or significant laboratory abnormalities, previously known or identified at screening, in the judgment of the investigator

Others:

* Pregnancy or breastfeeding or Women of childbearing age without effective contraception (a pregnancy test will be done)
* Subjects with excessive alcohol intake or drug abuse, in the judgment of the investigator
* Subjects who, in the opinion of the investigator, have a risk of non-compliance to the study procedures or who are otherwise not appropriate to include in this clinical trial (for example, being impossible to contact in case of emergency)

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects intended to participate will be recruited in Lille in the memory clinic and in the memory clinic network Meotis (North of France above Paris)
Sampling Method: Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2022-09-06 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Mean CSF-to-blood ratio (CBR) of leptin concentration. | At visit 2, occurring 1 to 90 days after visit 1(Baseline)
  Leptin concentration in blood and CSF (in the pg/mL range) will be measured by enzyme-linked immunosorbent assay (ELISA).

SECONDARY OUTCOMES:
Mean of the CSF-to-blood ratio (CBR) of hypothalamus-related hormones | At visit 2, occurring 1 to 90 days after visit 1(Baseline)
  CSF-to-blood ratio (CBR) of hypothalamus-related hormones
Blood metabolomics | At visit 2, occurring 1 to 90 days after visit 1(Baseline)
  Blood and CSF metabolites will be measured by LC MS/MS.Will be used a mix of targeted and untargeted approach for metabolomics using the Thermo Q-Exactive Orbitrap.
CSF metabolomics | At visit 2, occurring 1 to 90 days after visit 1(Baseline)
  Blood and CSF metabolites will be measured by LC MS/MS.Will be used a mix of targeted and untargeted approach for metabolomics using the Thermo Q-Exactive Orbitrap.
Correlation coefficient between leptin CBR and general cognitive functioning assessed by the Mattis Dementia Rating Scale (MDRS)6 | At visit 2, occurring 1 to 90 days after visit 1(Baseline)
  Correlation coefficient between leptin CBR and general cognitive functioning
Correlation coefficients between leptin CBR and performances in a neuropsychological battery assessing the function of affective and social cognition in each AD and FTD groups | At visit 2, occurring 1 to 90 days after visit 1(Baseline)
  Correlation coefficients between leptin CBR and performances
Correlation coefficients between leptin CBR and behavioral, and psychological symptoms of dementia | At visit 2, occurring 1 to 90 days after visit 1(Baseline)
  Correlation coefficients between leptin CBR and behavioral, and psychological symptoms
Correlation coefficients between leptin CBR and putative symptoms/markers of hypothalamus dysfunction | At visit 2, occurring 1 to 90 days after visit 1(Baseline)
  Correlation coefficients between leptin CBR and putative symptoms/markers
Correlation coefficients between leptin CBR and changes in resting metabolic activity assessed by indirect calorimetry through | At visit 2, occurring 1 to 90 days after visit 1(Baseline)
  Correlation coefficients between leptin CBR and changes in resting metabolic activity
Correlation coefficients between leptin CBR and the following CSF biomarkers | At visit 2, occurring 1 to 90 days after visit 1(Baseline)
  Correlation coefficients between leptin CBR and the following CSF biomarkers
Correlation coefficients between leptin CBR and the following MRI markers | At visit 2, occurring 1 to 90 days after visit 1(Baseline)
  Correlation coefficients between leptin CBR and the following MRI markers

CONTACTS AND LOCATIONS:
Overall Officials: Thibaud LEBOUVIER, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Memory Resources and Research Center Lille, Lille, France